CLINICAL TRIAL: NCT02344511
Title: A Phase 3, Multicenter, Double-Blind, Randomized, Comparator Controlled Trial of the Safety and Efficacy of Dalbavancin Versus Active Comparator in Pediatric Subjects With Acute Hematogenous Osteomyelitis of the Long Bones Known or Suspected to be Due to Gram-Positive Organisms
Brief Title: Dalbavancin vs Comparator in Pediatric Subjects With Acute Hematogenous Osteomyelitis
Acronym: AHOM
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Durata Therapeutics International BV (an Affiliate of Actavis, Inc.) (Industry)
Responsible Party: Sponsor
Organization: Durata Therapeutics Inc., an affiliate of Allergan plc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DUR001-304
Record Dates: First submitted 2015-01-10; First posted 2015-01-26 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Osteomyelitis
MeSH Terms: conditions — Osteomyelitis | interventions — dalbavancin; Cefazolin; Nafcillin; Oxacillin; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dalbavancin (Experimental): Patients with Creatine Clearance (CrCl) greater than 30 mL/min and patients receiving regular hemodialysis or peritoneal dialysis will receive 15 mg/kg Intravenous (IV) dalbavancin over 30 (+/- 5) minutes on Day 1 and on Day 8, not to exceed 1500 mg per administration in children at least 12 years and not to exceed 1000 mg per administration in children less than 12 years of age.
  • Patients with CrCl < 30 mL/min who are not receiving regular hemodialysis or peritoneal dialysis will receive 10 mg/kg IV dalbavancin over 30 (+/- 5) minutes on Day 1 and on Day 8, not to exceed 1000 mg per administration in children at least 12 years and not to exceed 750 mg per administration in children less than 12 years of age.
  Additionally, subjects randomized to the dalbavancin group will receive an IV placebo infusion at times corresponding to comparator group dosage times for the first eight days.
  Interventions: Drug: Dalbavancin
- 4 Comparators (Active Comparator): cefazolin, oxacillin, nafcillin or vancomycin according to the commercial label
  Patients with normal renal function will receive either vancomycin 15 mg/kg/dose, infused over 60 (+/- 10) minutes, every 6 hours (+/- 1 hour) not to exceed a daily total dose of 4000 mg, with dose adjustment based on local standard of care to achieve serum trough concentrations of 10 μg/mL to 20 μg/mL; or cefazolin 25 mg/kg/dose, infused over 60 (+/- 10) minutes, every 6 hours (+/- 1 hour); or nafcillin or oxacillin 50 mg/kg/dose, infused over 60 (+/- 10) minutes, every 6 hours (+/- 1 hour).
  Interventions: Drug: cefazolin, nafcillin, oxacillin or vancomycin

INTERVENTIONS:
Drug: Dalbavancin — Drug
  Other Names: Dalvance
  Arms: Dalbavancin
Drug: cefazolin, nafcillin, oxacillin or vancomycin — Standard of Care
  Arms: 4 Comparators

SUMMARY:
Dalbavancin for Pediatric Osteomyelitis

DETAILED DESCRIPTION:
A Phase 3, Multicenter, Double-Blind, Randomized, Comparator Controlled Trial of the Safety and Efficacy of Dalbavancin versus Active Comparator in Pediatric Subjects with Acute Hematogenous Osteomyelitis of the Long Bones Known or Suspected to be due to Gram-Positive Organisms.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 2-16 yrs
2. diagnosis of Acute Hematogenous Osteomyelitis (AHOM) of the long bones (ulna, radius, femur, tibia) defined by the following clinical signs and symptoms (< 2 weeks in duration; multiple sites of infection within long bones):
3. Limb abnormality: Pain, point tenderness upon palpation, motion restriction, loss of function
4. Magnetic resonance imaging (MRI) -OR- Gram-positive cocci documented on a Gram-stain from a bone specimen or from blood cultures.
5. Elevated C-Reactive Protein (CRP)
6. informed consent
7. willing and able to comply with the study protocol
8. Life Expectancy with appropriate antibiotic therapy and thru study duration

Exclusion Criteria:

1. Treatment with an investigational drug within 30 days preceding the first dose of study medication.
2. Receipt of > 24 hours of potentially effective intravenous antibacterial therapy for AHOM within 96 hours before randomization, unless the pathogen isolated was documented to be Methicillin resistant Staphylococcus aureus (MRSA) that was resistant to the administered antibiotic.
3. Evidence of subacute or chronic osteomyelitis including: symptoms > 2 weeks in duration
4. AHOM of non-long bones (e.g., pelvis or spine).
5. Extraosseous findings such as: subperiosteal abscess, pyomyositis, venous thrombosis, or pulmonary embolism.
6. Previous history of septic arthritis or osteomyelitis.
7. Major trauma, open-fracture, puncture wound of the foot, post-operative osteomyelitis, foreign body in or adjacent to affected bone or joint, or other iatrogenic bone or joint infections present at the site of infection.
8. Septic arthritis that is non-contiguous to osteomyelitis
9. Immunosuppression/immune deficiency
10. Evidence of Gram-negative bacteria by gram stain in the absence of Gram-positive organisms; fungus or mycobacteria at baseline.
11. Gram-negative bacteremia, even in the presence of gram-positive infection or gram-positive bacteremia.
12. A history of oral ulcers preceding the onset of musculoskeletal findings, recent gastrointestinal surgery (within 2 months)
13. Infection due to an organism known prior to study entry to be not susceptible to dalbavancin (dalbavancin mean inhibitory concentration > 0.12 µg/mL) or vancomycin (vancomycin mean inhibitory concentration (MIC) > 2 μg/mL).
14. Concomitant systemic antibacterial therapy for Gram-positive infections (eg. Rifampin, gentamicin).
15. Concomitant condition requiring any antibiotic therapy that would interfere with the assessment of study drug for the condition under study.
16. Sickle cell anemia.
17. Cystic fibrosis.
18. hypersensitivity to glycopeptide antibiotics.
19. not expected to survive for 3 months.
20. Positive urine (or serum) pregnancy test
21. Women of Child Bearing Potential who are unwilling or unable to use adequate contraceptive precautions.
22. Other severe acute or chronic medical or psychiatric condition would make the patient inappropriate for entry into this study.
23. Unwilling or unable to follow study procedures.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2018-10 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients with clinical improvement at Day 8 | Day 8

SECONDARY OUTCOMES:
Number of clinical responders | Day 8
Average reduction in C-reactive Protein (CRP) relative to the highest value | Day 8
Number of clinical responders by pathogen | Day 8
Number of Participants with Adverse Events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alena Jamdourek, MD, Study Director — Durata Therapeutics Inc., an affiliate of Allergan plc